CLINICAL TRIAL: NCT03109431
Title: Optimizing the HIV Treatment Continuum With a Stepped Care Model for Youth Living With HIV
Brief Title: Stepped Care for Youth Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Tulane University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Mary Jane Rotheram-Borus, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U19HD089886 - Study 2; U19HD089886 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: HIV; Mental Health; Illicit Substance Use; Sexually Transmitted Infections (STI)
Keywords: HIV Treatment Continuum; HIV Disease Progression; Mental Health; Substance Use; ARV Adherence; Retention in Care; STI
MeSH Terms: conditions — Psychological Well-Being; Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard Care (Experimental): Youth randomized to the Enhanced Standard Care arm will receive an Automated Messaging and Monitoring Intervention (AMMI), which involves receiving 1-5 texts per day to motivate, inform and refer to HIV care and health services. Message banks will focus on the HIV Treatment Continuum, with libraries dedicated to healthcare, wellness, sexual health, drug use and ARV adherence for YLH.
  Youth will also receive a weekly monitoring survey that covers six domains related to the HIV Treatment Continuum, including: ARV adherence, condomless sex, potential symptoms of STI, excessive use of alcohol and/or drugs, feelings of sadness or depression, and housing or food insecurity.
  Interventions: Behavioral: Level 1
- Stepped Care (Experimental): Youth randomized to the Stepped Care arm will receive up to three levels of intervention, depending on whether or not they have achieved viral suppression at each four-month assessment point. All youth will begin at Level 1 which is the same as the Enhanced Standard Care arm. If they fail to achieve viral suppression at a reassessment in four months, they will be moved to Level 2, which includes both Level 1 and enrollment in private, online peer support groups. If they fail to achieve viral suppression at another four-month assessment point, they will be moved to Level 3, which includes both Levels 1-2 and Coaching. Coaches will provide support using a strengths-based coaching approach.
  Interventions: Behavioral: Level 1; Behavioral: Level 2; Behavioral: Level 3

INTERVENTIONS:
Behavioral: Level 1 — Youth will receive 1-5 text messages per day for at least 12 months. Banks of about 750 messages (70-120 messages per domain) focus on the HIV Treatment Continuum, with messages focused on dedicated to healthcare, wellness, sexual health, drug use and medication reminders. Youth will be able to choose the time and frequency that they receive daily texts. Preferences for the timing and type of messages can be updated at 4-month assessment points.
  Youth will complete weekly monitoring surveys by text message. The survey will cover six domains related to the HIV Treatment Continuum. If YLH do not respond to the text, reminder messages will be sent to the youth. After three days of non-response a follow-up call by an interviewer will be made to the YLH.
Behavioral: Level 2 — Youth will be enrolled in online, private discussion groups.
  Peer Support will be offered by fellow participants and/or Youth Advisory Board members that have been trained in basic information on HIV, STI, drug use, mental health, homelessness, and stigma; using social media to create wall posts and use chat functions; and, how to initiate conversations on sensitive topics. By posting and responding to messages, Peer Supporters will encourage and broadly guide conversation related to the HIV Prevention Continuum, and other relevant topics.
  Coaches and Project Coordinators will be available to provide factual information (as needed), and remove inappropriate content.
  Arms: Stepped Care
Behavioral: Level 3 — Youth will have be assigned to a Coach trained in a strengths--based Coaching intervention, as well as common foundational theory, principles and skills used in adolescent HIV Evidence-Based Interventions (EBI). Youth preferences will drive the intervention delivery - whether in-person, electronically via the phone, email, text message, social media private messaging.
  Arms: Stepped Care

SUMMARY:
Optimizing the HIV Treatment Continuum with a Stepped Care Model for Youth Living with HIV (YLH) aims to achieve viral suppression among YLH. A cohort of 220 YLH will be identified in Los Angeles, CA and New Orleans, LA and recruited into a randomized controlled trial (RCT) with reassessments every 4 months over a 12 month follow-up period. The goal is to optimize the HIV Treatment Continuum over 12 months. YLH will be randomized into one of two study conditions: 1) Enhanced Standard Care Condition (n=110); or 2) Stepped Care (n=110). The Enhanced Standard Care condition will consist of an Automated Messaging and Monitoring Intervention (AMMI) with daily motivational, instructional and referral text messaging, and a brief weekly monitoring survey. The Stepped Care Condition will consist of three levels. Level 1 is the Enhanced Standard Care Condition. Level 2 is the Enhanced Standard Care Condition plus peer support using social media. Level 3 is the Enhanced Standard Care Condition and peer support plus coaching, which will be delivered primarily through electronic means (e.g., social media, text messaging, email, phone). All participants in the Stepped Care Condition begin at Level 1 but if they fail to have a suppressed viral load at any four-month assessment point, their intervention level will increase by one step until reaching Level 3.

DETAILED DESCRIPTION:
Viral suppression requires linkage and retention in care, as well as ARV adherence. These are key steps on the HIV Treatment Continuum. Youth Living with HIV (YLH) are far less likely to link or be retained in care, compared to adults. Only 36%-62% of YLH who know their serostatus are linked to medical care within 12 months of diagnosis. Young people are also more likely to drop out from care than adults 25+ years old. Among one sample was YLH (atypically 72% female), initial ARV adherence of 69%; but by one year, ARV adherence was negligible, because only 30% were retained in care. In one ATN study, of YLH, ARV adherence appeared to be about 50%. Originally an undetectable viral load was expected to require 95% ARV adherence. However rates as low as 70% may lead to viral suppression.

In this study, our primary outcome measure will be having a suppressed viral load (i.e., VL< 200) at each four month assessment for 12 months. Viral suppression typically requires adherence to ARV for 24 weeks until an undetectable viral load is achieved. There are many interpersonal and logistical barriers to retaining YLH in care and on ARV consistently. ARV adherence is related to the patient-provider relationship and to perceived side effects, the prescribed regimen, ease of getting ARV refills and a number of personal factors. Medication regimens are becoming much easier, as one pill a day is now one of the most highly used regimens. Unfortunately, the problem behaviors that lead to acquisition of HIV by YLH are factors which are consistently related to low adherence. Low adherence for both YLH and adults living with HIV is associated with younger age, depression, substance abuse and homelessness. Each of these challenges characterizes the lives of the YLH. The interventions proposed focus a great deal on problem-solving, automated messages, and monitoring of these comorbid conditions, so that ARV adherence is not derailed.

This study has a comprehensive retention plan to retain YLH. This plan will be particularly relevant to YLH nationally, who face challenges of homelessness, mental health problems, school-job issues, contact with criminal justice system and risks within their sexual partnerships, in addition to their seropositive HIV status. YLH are likely to deal with coming out as gay, bisexual or transgender, have substantial family conflict, to have abused drugs, may barter sex in order to survive and have a history of mental health problems or disorders. Studies of ARV adherence and retention in care have consistently found depression and the types of life challenges young people are experiencing to be directly related to engagement, retention and adherence to care over time. If the investigators fail to address these comorbid issues with YLH, they expect YLH to fail at achieving viral suppression.

Our Stepped Care approach aims to address these issues with increasingly intensive interventions, based on individual YLH's needs. While addressing comorbid issues may be more costly, it may have substantial saving in the YLH's lowered probability of transmitting HIV.

Stepped Care has been used as an intervention strategy with other chronic diseases and mental health disorders; the investigators believe this will be the first evaluation of stepped care with YLH. The Stepped Care model is a cost-effective and patient-centered approach for achieving better treatment outcomes for chronic illnesses. Under the Stepped Care model, simpler interventions are tried first with more intensive interventions reserved for those who do not benefit from the simple first-line treatments. Stepped Care might be an efficient method of delivering successfully more intensive interventions based on the YLH's behavior. If at any assessment (past a 12 month period when ARV initiated), a YLH in the Stepped Care condition demonstrates an unsuppressed viral load, the next level of intervention is triggered. The strategy typically makes best use of available resources for allocating resources to patients. Rather than everyone getting the same intervention, the dose and type of intervention is linked to outcomes.

An Automated Messaging and Monitoring (AMMI) is being proposed as the Enhanced Standard Care and the Level 1 of the Stepped Care Intervention. Both daily text messages, which aim to motivate, inform and encourage usage of care, and weekly probes regarding YLH's risk behaviors have been repeatedly linked to outcomes for a variety of conditions and populations. The investigators will tailor and adapt pre-existing libraries of theoretically-based messages that have been found successful in other RCTs with populations similar to this study - adults with HIV, transgender women, methamphetamine-using men who have sex with men (MSM) - for the YLH in this study. This is included with the Enhanced Standard Care condition as implementing an AMMI intervention is low-cost and easily scalable.

Level 2 of the Stepped Care Intervention will be electronically-based peer support, plus AMMI tailored to the YLH. Positive relationships are the second major dimension related to retention in care and adherence to ARV medications. Reviews of peer support among persons living with HIV, aimed at reducing stress, demonstrate peer support to be a critical intervention component. Peer support will be delivered through online, private social media groups. YLH will be incentivized to participate in online, private social media groups (i.e., posting and responding to topics) for period(s) of 4 months.

Peer Support will be offered by fellow participants and/or Youth Advisory Board members that have been trained in basic information on HIV, STI, drug use, mental health, homelessness, and stigma; using social media to create wall posts and use chat functions; and, how to initiate conversations on sensitive topics. By posting and responding to messages, Peer Supporters will encourage and broadly guide conversation related to the HIV Treatment Continuum, and other relevant topics. Coaches and Project Coordinators will be available to provide factual information (as needed), and remove inappropriate content.

Coaching - Level 3 - is the most intensive strategy for securing viral suppression and ARV adherence among YLH. Coaching has been used specifically to support families: to increase healthy eating and exercise, to enhance patient self-management and improve outcomes, to reduce community violence and domestic violence, to provide family therapy when some family members refuse, and to improve parenting skills around health and behavioral challenges. Now referred to as health coaching, these strategies differ from traditional health education by emphasizing goal-setting, problem-solving, and skill building. Coaching addresses multiple risk factors concurrently and aims to problem-solve emerging challenges.

This study will provide guidelines on how to implement Evidence-Based Practices, rather than replicating with fidelity an evidence-based intervention manual.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive serostatus
* Established HIV infection (not acutely infected)
* Able to provide informed consent

Exclusion Criteria:

* Youth under 12 years of age or above 24 years of age
* HIV-negative (high-risk HIV-negative youth will be invited to participate in another study)
* Acutely infected with HIV (RNA test will determine whether HIV infection is acute or established; acutely infected youth will be invited to participate in another study, once they are stable)
* Unable to understand the study procedures due to intoxication or cognitive difficulties (any youth who appear to be under the influence of alcohol or drugs will be unable to enroll in the study but invited to return at a later date)
* Unable to provide voluntary written informed consent

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Viral Suppression reflected as VL<200 | 12 month to 24 months
  Viral loads to be monitored at each 4-month assessment point using a blood draw and Quest Diagnostics HIV-1 quantitative real time-PCR in a research laboratory to measure HIV-1 RNA levels.

SECONDARY OUTCOMES:
Retention in Care | 12 month to 24 months
  At least two medical appointments annually, verified using medical charts
ARV Adherence | 12 month to 24 months
  Adherence is assumed through decreasing viral loads. Viral loads are assessed using Quest Diagnostics HIV-1 quantitative real time-PCR to measure HIV-1 RNA levels.
Reductions in Substance Use | 12 month to 24 months
  Rapid diagnostic tests (RDT) for alcohol, marijuana, methamphetamines, cocaine/crack, and opiates at each four-month assessment point
Sexual Partnerships | 12 month to 24 months
  Self-reported number of sexual partners, number of concurrent sexual partners, and condom use assessed at each four-month assessment point
Mental Health | 12 month to 24 months
  Self-reported symptoms of depression and anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Rotheram-Borus, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Tulane University Health Sciences Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zanoni BC, Mayer KH. The adolescent and young adult HIV cascade of care in the United States: exaggerated health disparities. AIDS Patient Care STDS. 2014 Mar;28(3):128-35. doi: 10.1089/apc.2013.0345. PMID 24601734
- [Background] Hall HI, Holtgrave DR, Maulsby C. HIV transmission rates from persons living with HIV who are aware and unaware of their infection. AIDS. 2012 Apr 24;26(7):893-6. doi: 10.1097/QAD.0b013e328351f73f. PMID 22313960
- [Background] Gardner JM, Powell CA, Baker-Henningham H, Walker SP, Cole TJ, Grantham-McGregor SM. Zinc supplementation and psychosocial stimulation: effects on the development of undernourished Jamaican children. Am J Clin Nutr. 2005 Aug;82(2):399-405. doi: 10.1093/ajcn.82.2.399. PMID 16087985
- [Background] Belzer ME, Fuchs DN, Luftman GS, Tucker DJ. Antiretroviral adherence issues among HIV-positive adolescents and young adults. J Adolesc Health. 1999 Nov;25(5):316-9. doi: 10.1016/s1054-139x(99)00052-x. PMID 10551660
- [Background] Ferrand R, Ford N, Kranzer K. Maximising the benefits of home-based HIV testing. Lancet HIV. 2015 Jan;2(1):e4-5. doi: 10.1016/S2352-3018(14)00039-3. Epub 2014 Dec 23. No abstract available. PMID 26424234
- [Background] Garofalo R, Kuhns LM, Hotton A, Johnson A, Muldoon A, Rice D. A Randomized Controlled Trial of Personalized Text Message Reminders to Promote Medication Adherence Among HIV-Positive Adolescents and Young Adults. AIDS Behav. 2016 May;20(5):1049-59. doi: 10.1007/s10461-015-1192-x. PMID 26362167
- [Background] Murphy DA, Belzer M, Durako SJ, Sarr M, Wilson CM, Muenz LR; Adolescent Medicine HIV/AIDS Research Network. Longitudinal antiretroviral adherence among adolescents infected with human immunodeficiency virus. Arch Pediatr Adolesc Med. 2005 Aug;159(8):764-70. doi: 10.1001/archpedi.159.8.764. PMID 16061785
- [Background] Fernandez MI, Huszti HC, Wilson PA, Kahana S, Nichols S, Gonin R, Xu J, Kapogiannis BG. Profiles of Risk Among HIV-Infected Youth in Clinic Settings. AIDS Behav. 2015 May;19(5):918-30. doi: 10.1007/s10461-014-0876-y. PMID 25117556
- [Background] Paterson DL, Swindells S, Mohr J, Brester M, Vergis EN, Squier C, Wagener MM, Singh N. Adherence to protease inhibitor therapy and outcomes in patients with HIV infection. Ann Intern Med. 2000 Jul 4;133(1):21-30. doi: 10.7326/0003-4819-133-1-200007040-00004. PMID 10877736
- [Background] Bangsberg DR. Less than 95% adherence to nonnucleoside reverse-transcriptase inhibitor therapy can lead to viral suppression. Clin Infect Dis. 2006 Oct 1;43(7):939-41. doi: 10.1086/507526. Epub 2006 Aug 23. PMID 16941380
- [Background] Murphy DA, Wilson CM, Durako SJ, Muenz LR, Belzer M; Adolescent Medicine HIV/AIDS Research Network. Antiretroviral medication adherence among the REACH HIV-infected adolescent cohort in the USA. AIDS Care. 2001 Feb;13(1):27-40. doi: 10.1080/09540120020018161. PMID 11177463
- [Background] Beach MC, Keruly J, Moore RD. Is the quality of the patient-provider relationship associated with better adherence and health outcomes for patients with HIV? J Gen Intern Med. 2006 Jun;21(6):661-5. doi: 10.1111/j.1525-1497.2006.00399.x. PMID 16808754
- [Background] Schneider J, Kaplan SH, Greenfield S, Li W, Wilson IB. Better physician-patient relationships are associated with higher reported adherence to antiretroviral therapy in patients with HIV infection. J Gen Intern Med. 2004 Nov;19(11):1096-103. doi: 10.1111/j.1525-1497.2004.30418.x. PMID 15566438
- [Background] Palepu A, Milloy MJ, Kerr T, Zhang R, Wood E. Homelessness and adherence to antiretroviral therapy among a cohort of HIV-infected injection drug users. J Urban Health. 2011 Jun;88(3):545-55. doi: 10.1007/s11524-011-9562-9. PMID 21409604
- [Background] Hudelson C, Cluver L. Factors associated with adherence to antiretroviral therapy among adolescents living with HIV/AIDS in low- and middle-income countries: a systematic review. AIDS Care. 2015;27(7):805-16. doi: 10.1080/09540121.2015.1011073. Epub 2015 Feb 23. PMID 25702789
- [Background] Greene JM, Ennett ST, Ringwalt CL. Prevalence and correlates of survival sex among runaway and homeless youth. Am J Public Health. 1999 Sep;89(9):1406-9. doi: 10.2105/ajph.89.9.1406. PMID 10474560
- [Background] Rice E, Barman-Adhikari A, Rhoades H, Winetrobe H, Fulginiti A, Astor R, Montoya J, Plant A, Kordic T. Homelessness experiences, sexual orientation, and sexual risk taking among high school students in Los Angeles. J Adolesc Health. 2013 Jun;52(6):773-8. doi: 10.1016/j.jadohealth.2012.11.011. Epub 2013 Jan 27. PMID 23360897
- [Background] Gonzalez JS, Batchelder AW, Psaros C, Safren SA. Depression and HIV/AIDS treatment nonadherence: a review and meta-analysis. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):181-7. doi: 10.1097/QAI.0b013e31822d490a. PMID 21857529
- [Background] Bower P, Gilbody S. Stepped care in psychological therapies: access, effectiveness and efficiency. Narrative literature review. Br J Psychiatry. 2005 Jan;186:11-7. doi: 10.1192/bjp.186.1.11. PMID 15630118
- [Background] Von Korff M, Tiemens B. Individualized stepped care of chronic illness. West J Med. 2000 Feb;172(2):133-7. doi: 10.1136/ewjm.172.2.133. No abstract available. PMID 10693379
- [Background] Zatzick D, Jurkovich G, Rivara FP, Russo J, Wagner A, Wang J, Dunn C, Lord SP, Petrie M, O'connor SS, Katon W. A randomized stepped care intervention trial targeting posttraumatic stress disorder for surgically hospitalized injury survivors. Ann Surg. 2013 Mar;257(3):390-9. doi: 10.1097/SLA.0b013e31826bc313. PMID 23222034
- [Background] Swendeman D, Ramanathan N, Baetscher L, Medich M, Scheffler A, Comulada WS, Estrin D. Smartphone self-monitoring to support self-management among people living with HIV: perceived benefits and theory of change from a mixed-methods randomized pilot study. J Acquir Immune Defic Syndr. 2015 May 1;69 Suppl 1(0 1):S80-91. doi: 10.1097/QAI.0000000000000570. PMID 25867783
- [Background] Swendeman D, Rotheram-Borus MJ. Innovation in sexually transmitted disease and HIV prevention: internet and mobile phone delivery vehicles for global diffusion. Curr Opin Psychiatry. 2010 Mar;23(2):139-44. doi: 10.1097/YCO.0b013e328336656a. PMID 20087189
- [Background] Swendeman D, Comulada WS, Ramanathan N, Lazar M, Estrin D. Reliability and validity of daily self-monitoring by smartphone application for health-related quality-of-life, antiretroviral adherence, substance use, and sexual behaviors among people living with HIV. AIDS Behav. 2015 Feb;19(2):330-40. doi: 10.1007/s10461-014-0923-8. PMID 25331266
- [Background] Swendeman D, Jana S, Ray P, Mindry D, Das M, Bhakta B. Development and Pilot Testing of Daily Interactive Voice Response (IVR) Calls to Support Antiretroviral Adherence in India: A Mixed-Methods Pilot Study. AIDS Behav. 2015 Jun;19 Suppl 2(0 2):142-55. doi: 10.1007/s10461-014-0983-9. PMID 25638037
- [Background] Yehia BR, Stewart L, Momplaisir F, Mody A, Holtzman CW, Jacobs LM, Hines J, Mounzer K, Glanz K, Metlay JP, Shea JA. Barriers and facilitators to patient retention in HIV care. BMC Infect Dis. 2015 Jun 28;15:246. doi: 10.1186/s12879-015-0990-0. PMID 26123158
- [Background] Rajabiun S, Mallinson RK, McCoy K, Coleman S, Drainoni ML, Rebholz C, Holbert T. "Getting me back on track": the role of outreach interventions in engaging and retaining people living with HIV/AIDS in medical care. AIDS Patient Care STDS. 2007;21 Suppl 1:S20-9. doi: 10.1089/apc.2007.9990. PMID 17563286
- [Background] Christopoulos KA, Massey AD, Lopez AM, Geng EH, Johnson MO, Pilcher CD, Fielding H, Dawson-Rose C. "Taking a half day at a time:" patient perspectives and the HIV engagement in care continuum. AIDS Patient Care STDS. 2013 Apr;27(4):223-30. doi: 10.1089/apc.2012.0418. PMID 23565926
- [Background] Rice E, Milburn NG, Rotheram-Borus MJ. Pro-social and problematic social network influences on HIV/AIDS risk behaviours among newly homeless youth in Los Angeles. AIDS Care. 2007 May;19(5):697-704. doi: 10.1080/09540120601087038. PMID 17505933
- [Background] Steinberg L, Morris AS. Adolescent development. Annu Rev Psychol. 2001;52:83-110. doi: 10.1146/annurev.psych.52.1.83. PMID 11148300
- [Background] Viner RM, Ozer EM, Denny S, Marmot M, Resnick M, Fatusi A, Currie C. Adolescence and the social determinants of health. Lancet. 2012 Apr 28;379(9826):1641-52. doi: 10.1016/S0140-6736(12)60149-4. Epub 2012 Apr 25. PMID 22538179
- [Background] Heimendinger J, Uyeki T, Andhara A, Marshall JA, Scarbro S, Belansky E, Crane L. Coaching process outcomes of a family visit nutrition and physical activity intervention. Health Educ Behav. 2007 Feb;34(1):71-89. doi: 10.1177/1090198105285620. Epub 2006 May 31. PMID 16740515
- [Background] Van Zandvoort M, Irwin JD, Morrow D. The impact of co-active life coaching on female university students with obesity. International Journal of Evidence Based Coaching and Mentoring. 2009;7(1):104-18.
- [Background] Kliewer W, Murrelle L, Prom E, Ramirez M, Obando P, Sandi L, Karenkeris MD. Violence exposure and drug use in central american youth: Family cohesion and parental monitoring as protective factors. Journal of Research on Adolescence. 2006;16(3):455-77.
- [Background] Huffman M. Health coaching: a new and exciting technique to enhance patient self-management and improve outcomes. Home Healthc Nurse. 2007 Apr;25(4):271-4; quiz 275-6. doi: 10.1097/01.NHH.0000267287.84952.8f. PMID 17426499
- [Background] Brown JL, Vanable PA. Cognitive-behavioral stress management interventions for persons living with HIV: a review and critique of the literature. Ann Behav Med. 2008 Feb;35(1):26-40. doi: 10.1007/s12160-007-9010-y. Epub 2008 Feb 16. PMID 18347902
- [Background] Salloum A, Robst J, Scheeringa MS, Cohen JA, Wang W, Murphy TK, Tolin DF, Storch EA. Step one within stepped care trauma-focused cognitive behavioral therapy for young children: a pilot study. Child Psychiatry Hum Dev. 2014 Feb;45(1):65-77. doi: 10.1007/s10578-013-0378-6. PMID 23584728
- [Background] Katz LF, Windecker-Nelson B. Domestic violence, emotion coaching, and child adjustment. J Fam Psychol. 2006 Mar;20(1):56-67. doi: 10.1037/0893-3200.20.1.56. PMID 16569090
- [Background] McGoldrick M, Carter B. Advances in coaching: family therapy with one person. J Marital Fam Ther. 2001 Jul;27(3):281-300. doi: 10.1111/j.1752-0606.2001.tb00325.x. PMID 11436422
- [Background] Mabe PA, Turner MK, Josephson AM. Parent management training. Child Adolesc Psychiatr Clin N Am. 2001 Jul;10(3):451-64. PMID 11449806
- [Background] Morawska A, Stallman HM, Sanders MR, Ralph A. Self-directed behavioral family intervention: Do therapists matter? Child & Family Behavior Therapy. 2005;27(4):51-72.
- [Background] Butterworth S, Linden A, McClay W. Health Coaching as an Intervention in Health Management Programs. Disease Management and Health Outcomes. 2007;15(5):299-307.
- [Background] Merson MH, O'Malley J, Serwadda D, Apisuk C. The history and challenge of HIV prevention. Lancet. 2008 Aug 9;372(9637):475-88. doi: 10.1016/S0140-6736(08)60884-3. Epub 2008 Aug 5. PMID 18687461
- [Background] Ooms G, Van Damme W, Baker BK, Zeitz P, Schrecker T. The 'diagonal' approach to Global Fund financing: a cure for the broader malaise of health systems? Global Health. 2008 Mar 25;4:6. doi: 10.1186/1744-8603-4-6. PMID 18364048
- [Background] Rotheram-Borus MJ, Swendeman D, Flannery D, Rice E, Adamson DM, Ingram B. Common factors in effective HIV prevention programs. AIDS Behav. 2009 Jun;13(3):399-408. doi: 10.1007/s10461-008-9464-3. Epub 2008 Oct 2. PMID 18830813
- [Derived] Arnold EM, Kamal S, Rotheram-Borus MJ, Bridges SK, Gertsch W, Norwood P, Swendeman D; Adolescent Medicine Trials Network (ATN) CARES Team. Factors Associated With Antiretroviral Adherence Among Youth Living With HIV. J Acquir Immune Defic Syndr. 2024 Mar 1;95(3):215-221. doi: 10.1097/QAI.0000000000003345. PMID 37977178
- [Derived] Arnold EM, Yalch MM, Christodoulou J, Murphy DA, Swendeman D, Rotheram-Borus MJ; Adolescent Medicine Trials Network CARES Study Team. Rumination influences the relationship between trauma and depression over time among youth living with HIV. J Affect Disord. 2023 Feb 1;322:9-14. doi: 10.1016/j.jad.2022.11.010. Epub 2022 Nov 9. PMID 36370915
- [Derived] Arnold EM, Swendeman D, Harris D, Fournier J, Kozina L, Abdalian S, Rotheram MJ; Adolescent Medicine Trials Network CARES Team. The Stepped Care Intervention to Suppress Viral Load in Youth Living With HIV: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Feb 27;8(2):e10791. doi: 10.2196/10791. PMID 30810536
- See also: AIDS Action Committee. (2015). Adolescents, young adults & the HIV/AIDS continuum. — http://www.aac.org